CLINICAL TRIAL: NCT04546945
Title: Resident Doctor at Clinical Pathology Department
Brief Title: Aberrant Expression of CD56 in Patients With Hematologic Malignancies.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asmaa Hassan mohamed Abdel Mawjoud (Other)
Responsible Party: Sponsor-Investigator, Asmaa Hassan mohamed Abdel Mawjoud, resident doctor clinical pathology, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Asmaa Hassan
Record Dates: First submitted 2020-09-03; First posted 2020-09-14 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control cases: normal healthy person
  Interventions: Diagnostic Test: CD56
- Patients: Patients with hematologic malignancies. Newly diagnosed.
  Interventions: Diagnostic Test: CD56

INTERVENTIONS:
Diagnostic Test: CD56 — detection of CD56 by flow cytometry

SUMMARY:
CD56(cluster of differentiation 56) was found to be ectopically expressed in multiple myeloma . A met analysis indicated that CD56 over expression may be an adverse prognostic factor in AML. To the best of our knowledge, no available data the expression pattern of CD56 in other Hematologic malignancies. This work is designed to evaluate the expression pattern of CD56 in hematologic malignancies.

DETAILED DESCRIPTION:
CD56 is the archetypal phenotypic marker of natural killer cells but can actually be expressed by many more immune cells, including alpha, beta T cells, gamma, delta T cells, dendritic cells, and monocytes. Common to all these CD56 expressing cell types have strong immunostimulatory effector functions, including T helper 1 cytokine production and an efficient cytotoxic capacity. Interestingly, both numerical , functional deficiencies and phenotypic alterations of the CD56 immune cell fraction have been reported in patients with various infectious, autoimmune, or malignant diseases.CD56 is also known as neural cell adhesion molecule (NCAM).

Hematologic malignancies are a heterogeneous group of diseases of diverse incidence, prognosis and etiology that arise from malignant transformation of cells from the bone marrow or the lymphatic system.There are two major groups of Hematologic malignancies according to their cell lineage: Myeloid and lymphoid. Lymphoid neoplasms are a varied group that includes non-Hodgkin lymphoma (NHL), Hodgkin lymphoma (HL), leukemia and multiple myeloma (MM).myeloid neoplasms and acute leukaemia include: Myeloproliferative neoplasms (MPN), Myelodysplastic/myeloproliferative neoplasms (MDS/MPN), Myelodysplastic syndromes (MDS), Acute myeloid leukaemia (AML), Acute leukemias of ambiguous lineage, B-lymphoblastic leukaemia/lymphoma, T-lymphoblastic leukaemia/lymphoma.The exact causes of Hematologic malignancies are still unknown although multiple epidemiological studies have reported an association between the development of Hematologic malignancies and several risk factors. Some factors are well documented to increase the risk of some types of leukaemia such as benzene exposure and ionizing radiation.However, many other factors were observed to have an association with Hematologic malignancies such as age, gender, tobacco smoking , obesity , hepatitis C virus (HCV) infection , family history , and environmental exposure to pesticides but with no clear evidence.

CD56 was found to be ectopically expressed in multiple myeloma. A met analysis indicated that CD56 over expression may be an adverse prognostic factor in AML. To the best of our knowledge, no available data the expression pattern of CD56 in other Hematologic malignancies. This work is designed to evaluate the expression pattern of CD56 in hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies.
* Newly diagnosed

Exclusion Criteria:

* Patients with hematologic disorders other than hematologic malignancies.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hematologic malignancies Newly diagnosed
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
To identify the Pattern of expression of CD56 in hematologic malignancies. | 1 years
  Expression of aberrant CD56 in hematologic malignancies by flowcytometry. To explore incidence of Expression of aberrant CD56 in hematologic malignancies .
  Correlation between this expression and outcome of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Maged S Mahmoud, prof, Study Director — Assiut University
Locations (2):
- Egypt (2):
  - Assiut University, Asyut
  - Assiut university, Asyut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: (1) Kelly-Rogers J, Madrigal-Estebas L, O'Connor T, Doherty DG. Activation-induced expression of CD56 by T cells is associated with a reprogramming of cytolytic activity and cytokine secretion profile in vitro. Hum Immunol (2006) — https://www.google.com/search?q=Kelly-Rogers+J%2C+Madrigal-Estebas+L%2C+O%E2%80%99Connor+T%2C+Doherty+DG.+Activation-induced+expression+of+CD56+by+T+cells+is+associated+with+a+reprogramming+of+cytolytic+activity+and+cytokine+secretion+profile+in+vitro.+Hum+Immunol+(2006)&oq=Kelly-Rogers+J%2C+Madrigal-Estebas+L%2C+O%E2%80%99Connor+T%2C+Doherty+DG.+Activation-induced+expression+of+CD56+by+T+cells+is+associated+with+a+reprogramming+of+cytolytic+activity+and+cytokine+secretion+profile+in+vitro.+Hum+Immunol+(2006)+&aqs=chrome..69i57.1761j0j15&sourceid=chrome&ie=UTF-8
- See also: Roothans D, Smits E, Lion E, Tel J, Anguille S. CD56 marks human dendritic cell subsets with cytotoxic potential. Oncoimmunology (2013) — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3601173/
- See also: (3) Van Acker HH, Anguille S, Willemen Y, Van den Bergh JM, Berneman ZN, Lion E, et al. Interleukin-15 enhances the proliferation, stimulatory phenotype, and antitumor effector functions of human gamma delta T cells. J Hematol Oncol (2016) — https://pubmed.ncbi.nlm.nih.gov/27686372/
- See also: Heleen H. Van Acker,* Anna Capsomidis, Evelien L. Smits, and Viggo F. Van Tendeloo ( CD56 in the Immune System: More Than a Marker for Cytotoxicity?) Published 2017 frontiers in immunology. — https://www.frontiersin.org/articles/10.3389/fimmu.2017.00892/full
- See also: (6) Sant M, Allemani C, Tereanu C, De Angelis R, Capocaccia R, Visser O, Marcos-Gragera R, Maynadie M, Simonetti A, Lutz JM, et al: Incidence of hematologic malignancies in Europe by morphologic subtype: Results of the HAEMACARE project. Blood. — https://pubmed.ncbi.nlm.nih.gov/20664057/
- See also: (8)Vardiman JW, Thiele J, Arber DA, Brunning RD, Borowitz MJ, Porwit A, Harris NL, Le Beau MM, Hellström-Lindberg E, Tefferi A and Bloomfield CD: The 2008 revision of the World Health Organization (WHO) — https://pubmed.ncbi.nlm.nih.gov/19357394/
- See also: (9) Swerdlow SH, Campo E, Pileri SA, Harris NL, Stein H, Siebert R, Advani R, Ghielmini M, Salles GA, Zelenetz AD and Jaffe ES: The 2016 revision of the World Health Organization classification of lymphoid neoplasmsBlood. — https://pubmed.ncbi.nlm.nih.gov/26980727/
- See also: (10) A. Arber, Attilio Orazi,Hasserjian, J ¨urgen Thiele,J. Borowitz,Le Beau, D. Bloomfield, Cazzola, and W. Vardiman : The 2016 revision to the World Health Organization classification of myeloid neo — https://pubmed.ncbi.nlm.nih.gov/27069254/
- See also: (11) Rodriguez-Abreu D, Bordoni A, Zucca E. Epidemiology of hematological malignancies. Ann Oncol 2007. — https://pubmed.ncbi.nlm.nih.gov/17311819/
- See also: (12) Floderus B, Persson T, Stenlund C, Wennberg A, Ost A, Knave B. Occupational exposure to electromagnetic fields in relation to leukemia and brain tumors: a case-control study in Sweden. Cancer Causes Control 1993 — https://pubmed.ncbi.nlm.nih.gov/8218879/
- See also: (13) Kedia S, Bhatt VR, Rajan SK, Tandra PK, El Behery RA, Akhtari M. Benign and malignant hematological manifestations of chronic hepatitis C virus infection. Int J Prev Med 2014. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4635414/
- See also: (14) Pan Y, Wang H, Tao Q, Zhang C, Yang D, Qin H, et al. Absence of both CD56 and CD117 expression on malignant plasma cells is related with a poor prognosis in patients with newly diagnosed multiple myeloma. Leuk Res (2016) — https://pubmed.ncbi.nlm.nih.gov/26597998/
- See also: (15) Xu S, Li X, Zhang J, Chen J. Prognostic value of CD56 in patients with acute myeloid leukemia: a meta-analysis. J Cancer Res Clin Oncol (2015) — https://pubmed.ncbi.nlm.nih.gov/25924702/
- See also: (16) Hazra A. Using the confidence interval confidently. J Thorac Dis 2017. — http://jtd.amegroups.com/article/view/16406/html